CLINICAL TRIAL: NCT02104388
Title: A Double-Masked, Randomized, Multicenter, Placebo-Controlled, Parallel-Group Study of SJP-0035 Ophthalmic Solution Compared With Placebo to Assess Safety and Efficacy of SJP-0035 Ophthalmic Solution for Corneal Epithelial Wound Healing in Patients With Moderate to Severe Corneal Epithelial Disorders
Brief Title: Safety and Efficacy Study of SJP-0035 Ophthalmic Solution in Patients With Moderate to Severe Corneal Epithelial Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Senju Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJP-0035/2-01
Record Dates: First submitted 2014-03-19; First posted 2014-04-04 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Corneal Epithelial Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SJP-0035 Ophthalmic Solution (Experimental): Patients randomized to the SJP-0035 Ophthalmic solution will receive 1 drop in the affected eye(s) given 4 times daily for 4 weeks.
  Interventions: Drug: SJP-0035 Ophthalmic Solution
- Vehicle of SJP-0035 Ophthalmic Solution (Placebo Comparator): Patients randomized to the placebo arm will receive 1 drop in the affected eye(s) given 4 times daily for 4 weeks.
  Interventions: Drug: Vehicle of SJP-0035 Ophthalmic Solution

INTERVENTIONS:
Drug: SJP-0035 Ophthalmic Solution
  Arms: SJP-0035 Ophthalmic Solution
Drug: Vehicle of SJP-0035 Ophthalmic Solution
  Arms: Vehicle of SJP-0035 Ophthalmic Solution

SUMMARY:
The purpose of the study is to determine if SJP-0035 ophthalmic solution is effective in promoting corneal epithelial wound healing in conditions associated with corneal epithelial disorders.

DETAILED DESCRIPTION:
There is currently no product approved for corneal epithelial wound healing. A Phase 1 Study SJP-0035/1-01 was conducted in healthy volunteers to investigate the safety, tolerability, and pharmacokinetic profile of SJP-0035 ophthalmic solution and to determine the appropriate dose to be evaluated in patients with moderate to severe corneal epithelial disorders.

This Phase 2a study is being conducted to evaluate the safety and efficacy of SJP-0035 ophthalmic solution in patients to promote corneal epithelial wound healing in conditions associated with corneal epithelial disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 75 years, inclusive.
* Has moderate to severe superficial punctate keratitis (SPK) and/or corneal erosion in 1 or both eyes.
* Has symptoms caused by corneal epithelial disorders.
* Has not obtained improvement from previous treatment for the SPK or corneal erosion within the last 30 days.
* Is a female of childbearing potential with a negative pregnancy test result at Screening and baseline and agrees to use effective contraception throughout the study or is a postmenopausal woman with a negative pregnancy test result at Screening and baseline.

Exclusion Criteria:

* Has any corneal stromal or endothelial abnormalities including an active bacterial or viral ocular infection, bullous keratopathy, or chemical burns or any trauma to the cornea.
* Any active or chronic allergic, bacterial, or viral infection of ocular adnexa and eye structures.
* Had previous ocular/refractive surgery (including laser surgery) within the last 6 months.
* Has used any ocular medication (except mydriatics, stain, and topical anesthesia used for study assessments) within 14 days prior to the first dose of study drug, or who are anticipated to require such medications during the study. Artificial tears may be used up to 72 hours prior to the first dose.
* Is unable to discontinue Restasis. A 28-day washout period prior to the first dose of study drug is required.
* Is a contact lens wearer and cannot discontinue use for the duration of the study.
* Alcohol or drug abuse within the past 6 months.
* Positive hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus test at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2015-08-04 (Actual); Study Completion 2015-08-04 (Actual)

PRIMARY OUTCOMES:
Clearing of corneal fluorescein staining at week 4 | measured at Week 4
  A patient will be considered a success for clearing of corneal fluorescein staining if their fluorescein staining has disappeared.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety. | baseline up to week 18
  An Adverse Event is defined as any untoward medical occurrence in a patient enrolled into the study regardless of its causal relationship to study drug.
Changes of subjective symptoms: blurred vision, photophobia and eye irritation | screening up to week 18
  100-point assessments are performed for the symptom of blurred vision, photophobia and eye irritation.
Changes of subjective signs: tear stability, conjunctival epithelia, and surface curvature of cornea | screening up to week 18
  These changes are measured at every study visit using standard ophthalmology procedures.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Senju Investigational Site, Little Rock, Arkansas
  - Senju Investigational Site, Glendale, California
  - Senju Investigational Site, Glendora, California
  - Senju Investigational Site, Huntington Beach, California
  - Senju Investigational Site, Lancaster, California
  - Senju Investigational Site, Newport Beach, California
  - Senju Investigational Site, Pasadena, California
  - Senju Investigational Site, Petaluma, California
  - Senju Investigational Site, Santa Maria, California
  - Senju Investigational Site, Hoffman Estates, Illinois
  - Senju Investigational site, Edgewood, Kentucky
  - Senju Investigational Site, Kansas City, Missouri
  - Senju Investigational Site, Palisades Park, New Jersey
  - Senju Investiational Site, Rochester, New York
  - Senju Investigational Site, High Point, North Carolina
  - Senju Investigational Site, Rapid City, South Dakota
  - Senju Investigational Site, Norfolk, Virginia